CLINICAL TRIAL: NCT05500027
Title: The Diagnostic and Survival Predictive Value of Peripheral Serum Soluble CD58 (sCD5858) in Pancreatic Cancer Patients
Brief Title: sCD8, as a Novel Biomarker for Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiaofei Liu, Department of General Surgery, Peking Union Medical College Hospital
Other Study IDs: JS-2954
Record Dates: First submitted 2022-08-07; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Serum Biomarker; Pancreatic Cancer
Keywords: CD58; TGFβ1; Serum biomaker; Pancreatic cancer; Early dection
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Pancreatic cancer: All TNM stages of pancreatic cancer, before/after surgery, before/after chemotherapy, before/after bile drainage
  Interventions: Diagnostic Test: serum test
- Low malignant grade of pancreatic neoplasms: IPMN, MCN, PNEN, and SPN
  Interventions: Diagnostic Test: serum test
- Pancreatitis: acute, chronic, and auto-immune pancreatitis
  Interventions: Diagnostic Test: serum test
- Auto-immune diseases: SLE, RA, et al
  Interventions: Diagnostic Test: serum test
- Pancreatic-biliary infections: cholecystitis, cholangitis, et al
  Interventions: Diagnostic Test: serum test

INTERVENTIONS:
Diagnostic Test: serum test — serum test of sCD58 and TGFbeta1

SUMMARY:
Early detection and early treatment is the most important issue to improve the long-term survival of pancreatic cancer patients. CA199 is the most commonly used biomarker for early detection and to predict survival, however, the overall positive rate for CA199 is only 75%, and what is worse, for the early stage of pancreatic cancer patients, the positive rate is even lower, and for the lewis negative patients, CA199 is not produced at all. Therefore, novel biomarkers for the early detection of pancreatic cancer are still urgently needed. Previously, we found there is a vicious cycle between pancreatic cancer cells, that is pancreatic cancer-produced TGFbeta1 could promote the production of soluble CD58 (sCD58) in macrophages, and then sCD58 could induce the production of TGFbeta1 in pancreatic cancer cells. Therefore, the serum level of TGFbeta1 and sCD58 has diagnostic and survival values for pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly malignant tumor with a very poor prognosis. The five-year survival rate is only 10%, and its incidence is significantly increasing worldwide. Early diagnosis and treatment can improve the survival of pancreatic cancer patients. However, the early diagnosis of pancreatic cancer is extremely difficult, and more than 50% of patients have distant metastasis at the time of diagnosis. Therefore, the development of sensitive and efficient serum biomarkers for pancreatic cancer has important clinical significance. Pancreatic cancer has a special microenvironment. Pancreatic cancer cells are only 10 to 30 percent, while inflammatory cells are more than 50 percent. The interaction between inflammatory cells and tumor cells promotes the development of pancreatic cancer. CD58 is an important immune adhesion molecule, which exists in the membrane (mCD58) and soluble (sCD58) states. For the first time, the investigators found that macrophages can promote CD58 expression separation in pancreatic cancer cells through TGFβ1, that is, the expression of mCD58 decreased and the release of more sCD58. SCD58 competitively binds CD2 on T/NK cells, thereby inducing immune suppression and promoting the development of pancreatic cancer. Therefore, the investigators propose a scientific hypothesis that serum sCD58 and TGFβ1 can be used as markers of tumor burden and tumor immunosuppression status in pancreatic cancer. They have important value in the diagnosis, immunotyping, and prognosis of pancreatic cancer. To test this scientific hypothesis, the investigators obtained peripheral blood serum from 132 healthy controls, 131 patients undergoing pancreatic cancer surgery, 80 patients with low-grade malignant pancreatic tumors, 58 patients with benign pancreatic tumors, and 16 patients with chronic pancreatitis as a training cohort. The expression levels of sCD58 and TGFβ1 in serum were detected by Elisa. The results showed that the expression levels of sCD58 and TGFβ1 in peripheral blood were significantly higher in pancreatic cancer, but there was no significant difference in sCD58 and TGFβ1 between other pancreatic diseases and healthy people. The expression levels of sCD58 and TGFβ1 were positively correlated with the clinical stage of pancreatic cancer. The level of sCD58 is negatively correlated with the prognosis of pancreatic cancer patients. The three-factor diagnostic model of sCD58, TGFβ1 and CA199 can improve the diagnostic efficiency of pancreatic cancer, especially when CA199 is disabled, sCD58 and TGFβ1 still have high diagnostic efficiency. However, this previous study still had the following shortcomings :(1) patients with advanced pancreatic cancer were not included; (2) The relationship between serum sCD58 and TGFβ1 and the efficacy of chemotherapy was not clarified. (3) The effects of immune diseases and infection on serum sCD58 and TGFβ1 were not considered; (4) The included sample size is small. Based on the previous study, this study plans to expand the sample size by 2 times as the validation cohort. The clinical value of serum sCD58 and TGFβ1 as biomarkers for diagnosis, immunotyping and prognosis prediction of pancreatic cancer was fully clarified by using pre-mature detection methods and modeling methods to improve the above four deficiencies. To develop a kit combining sCD58, TGFβ1 and CA199, improve the early diagnosis and treatment rate of pancreatic cancer, guide accurate immune typing and optimize individualized treatment, and finally prolong the survival time of patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Stage I-IV pancreatic cancer patients with pathological diagnosis
* Pancreatic cancer patients before and 1 week after surgery
* Pancreatic cancer patients before and 1 week after bile drainage
* IPMN patients with pathological diagnosis before and 1 week after surgery
* MCN patients with pathological diagnosis before and 1 week after surgery
* SPN patients with pathological diagnosis before and 1 week after surgery
* PNEN patients with pathological diagnosis before and 1 week after surgery
* Chronic pancreatitis patients with pathological diagnosis
* Cholecystitis patients meeting clinical criteria
* Cholangitis patients meeting clinical criteria
* Autoimmune diseases meeting clinical criteria

Exclusion Criteria:

* Refusal to participate
* Age less than 18-year old and over 85-year old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A pathological diagnosis should be obtained for cancer patients. In addition, the other non-neoplastic disease patients should reach the diagnostic criteria recommended by the related guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differentiation expression of serum sCD58 and TGfbeta1 among pancreatic cancer and other conditions | 4 years
  Serum sCD58 and TGFbeta1, alone or in combination with CA19-9, has diagnostic and survival predictive value for pancreatic cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Qiaofei Liu, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Liu Q, Yang S, Liao Q. CD58 Immunobiology at a Glance. Front Immunol. 2021 Jun 8;12:705260. doi: 10.3389/fimmu.2021.705260. eCollection 2021. PMID 34168659
- [Result] Zhang Y, Liu Q, Liu J, Liao Q. Upregulated CD58 is associated with clinicopathological characteristics and poor prognosis of patients with pancreatic ductal adenocarcinoma. Cancer Cell Int. 2021 Jun 30;21(1):327. doi: 10.1186/s12935-021-02037-0. PMID 34193136